CLINICAL TRIAL: NCT06095752
Title: Spectrum of Blood Viscosity , Albumin / Fibrinogen Ratio and Red Cell Distribution Width in Newly Diagnosed Multiple Myeloma Patients. Observation Study
Brief Title: Multiple Myeloma Prognostic Indices
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Radwan Abdelhakim, Resident doctor, Ahmed Radwan abdelhakim, Assiut University
Other Study IDs: MM prognosis
Record Dates: First submitted 2023-09-27; First posted 2023-10-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma; Hematologic Diseases
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases | interventions — Blood Viscosity; Albumins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: blood viscosity , albumin / fibrinogen ratio and red cell distribution — In multiple myeloma patients ,we get blood viscosity , albumin / fibrinogen ratio and red cell distribution directly after confirmed diagnosis to determine the prognosis of the disease in association with these tests results

SUMMARY:
The aim of this study was to evaluate the impact of albumin / fibrinogen ratio, blood viscosity and RDW on the prognosis of a newly diagnosed MM patients

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a hematologic neoplasm of plasma cells that arises in the bone marrow, manifest by bone pain, pathologic fractures, anemia, renal insufficiency and recurrent infections. Treatment options include chemotherapy (proteosome inhibitors), targeted therapy, autologous stem cell transplantation and supportive care. MM has numerous prognostic factors affecting patient outcomes, some of the most important prognostic factors include age, stage of disease, levels of certain proteins like Beta -2 microglobulin, albumin, chromosomal abnormalities and renal function tests. In addition to albumin / fibrinogen ratio, blood viscosity and hematologic indices which are mainly focused on through this research .

The albumin / fibrinogen ratio has been recently studied as a potential prognostic factor for newly diagnosed MM patients, fibrinogen is the protein that plays a role in blood clotting, while albumin helps regulate fluid balance in the body. Studies show that a higher albumin/ fibrinogen ratio is associated with a better prognosis of MM, However, further studies is necessary to fully understand the impact of this ratio on MM prognosis.

Blood viscosity is the measure of the thickness and stickiness of the blood, which can impact blood flow and oxygen delivery to vital organs. Newly diagnosed MM patients, higher whole blood viscosity is associated with a poorer prognosis and shorter survival times. increased viscosity may contribute to the development of blood clots and impaired circulation, leading to tissue damage and organ failure, However, further studies is needed to better understand the mechanism underlying this relationship and develop targeted interventions to improve outcomes.

Several studies have shown that radial distribution width (RDW) can serve as a prognostic factor in the newly diagnosed MM patients. This index can provide important information about patients' immune response, inflammation and overall health status. A high RDW are associated with poor prognosis. However, further studies is necessary to fully understand the impact of these indices on MM prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with MM according to International Myeloma Working Group criteria 2016.

Exclusion Criteria:

* Patient previously diagnosed MM and started treatment or in post treatment follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: based on study methodology , the studied population (who are the newly diagnosed cases ) will be followed up to one year after diagnosis to report outcomes . the researcher will recruit the newly diagnosed cases who seek care at internal medicine department, assiut university hospital in completed one year duration and then follow up the case for one year. After reviewing medical record , average flow rate of MM at internal medicine department is 2 cases per month , nearly 25 cases will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Determine the prognosis of newly diagnosed multiple myeloma patients in survival for one year. | One year
  After initial diagnosis of a patient to have multiple myeloma , blood viscosity is obtained and within a year , a relation is established between the prognosis of the disease and the initial results of blood viscosity
Determine the prognosis of newly diagnosed multiple myeloma patients in survival for one year. | One year
  After initial diagnosis of a patient to have multiple myeloma , albumin / fibrinogen ratio is obtained and within a year , a relation is established between the prognosis of the disease and the initial results of albumin /fibrinogen ratio
Determine the prognosis of newly diagnosed multiple myeloma patients in survival for one year. | One year
  After initial diagnosis of a patient to have multiple myeloma , red cell distribution is obtained and within a year , a relation is established between the prognosis of the disease and the initial results of red cell distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt